CLINICAL TRIAL: NCT03199729
Title: Aging and Mixed Perturbation Training to Reduce Falls in Locomotion
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Tanvi Bhatt, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0887; 1R01AG050672-01A1 (NIH)
Record Dates: First submitted 2017-06-19; First posted 2017-06-27 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Older Adults
Keywords: Overground training; Dynamic Stability; Fall risk

STUDY DESIGN:
Intervention Model Description: Controlled design to understand the mechanisms of adaptive interference and generalization, their interaction with retention, and how these can be applied to maximize training effects for minimizing falls-risk among older adults.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Slip-only training (Experimental): Overground, slip specific perturbation training only delivered in a fixed sequence. After the baseline walking trials, subjects will walk for 30-35 trials, after which training will begin consisting of a first block of 8 repeated slips (S1-S8), a block of 3 regular (non-perturbed) walking trials (W1-W3), another block of 8 slips (S9-16), a second block of 3 regular walking trials (W4-W6), and a final block of 8 slips (S17-S24) mixed with 10 regular walking trials.
  Interventions: Other: Slip-only training
- Trip-only training (Experimental): Trip specific training delivered in an identical sequence (mixed with non-trip trials) as the Group with slip only training.
  Interventions: Other: Trip-only training
- Control (No Intervention): Walk for about 70-75 trials at the preferred walking pace to match the total trials the other groups receive before the test perturbations.
- Combined slip+trip training (Experimental): Training consisting of repeated exposure to both slips and trips.
  Interventions: Other: Combined slip+trip training

INTERVENTIONS:
Other: Slip-only training — Subjects in this arm will receive overground, slip specific perturbation training only. The total perturbation training trials received by this group will be 24 but the protocol will consist of a total of 70-75 trials (to match the training length and time of Combined slip and trip training group).
  Arms: Slip-only training
Other: Trip-only training — Subjects in this arm consisting of a total of 24 trials of trip specific training delivered in an identical sequence (mixed with non-trip trials) as the Group with slip only training.
  Arms: Trip-only training
Other: Combined slip+trip training — Subjects in this arm will receive training consisting of repeated exposure to both slips and trips with a total of 24 slips plus 24 trips to keep the number of trials of each perturbation same as the perturbation specific training groups (slip only and trip only), however, the total dose will be doubled. The total trials walked (perturbed + unperturbed) will be 75.
  Arms: Combined slip+trip training

SUMMARY:
The long-term objective of this research is to develop an efficacious training paradigm to enhance older adults' defense mechanisms against falls and possibility reduce healthcare cost. The Centers for Disease Control and Prevention estimates the direct medical cost for fall related injuries to be $30 billion annually. Slips and trips combined account for more than 50% of the outdoor falls in community-dwelling older adults. These environmental perturbations are opposing in nature, with slips mainly resulting in backward falls and trips in forward falls. This project explores perturbation training through both slip and trip exposure based on the principles of motor learning. The project design consists of a randomized controlled trial to examine the ability of the central nervous system to mitigate the interference in stability control (if any) that is induced by opposing types of perturbations. It also introduces a novel combined slip and trip perturbation training paradigm to enhance one's ability to retain and generalize the acquired fall-prevention skills to both types of falls. Slips and trips induced on an over ground walkway will be used to prepare the motor system to improve stability control and vertical limb support to resist falls. The longer-term benefits of such combined perturbation training over exclusive slip-only or trip-only perturbation training in reducing both laboratory-induced and real life falls will also be assessed. The hypothesis of this study if supported by the results will provide an evidence-supported training protocol to reduce the fall-risk among community-dwelling older adults.

DETAILED DESCRIPTION:
Impaired or delayed reactive postural responses pose a potential threat to falls while walking resulting in slips or trips in older and neurologically impaired individuals. Therefore, increase in understanding of postural responses to unexpected external perturbation in older adults and people with neurological diseases will lead to development of new therapeutic approaches for fall prevention in this population. The overall objective of this is to investigate the dynamic stability during slip and trip-like experiences by evaluating the efficiency of recovery responses, retention and fall-risk reduction to slips or trips induced during normal walking in healthy older adults. Participants will be community dwelling ambulatory older adults between the age range of 60 to 90 years. Subjects will be screened for the inclusion criteria. Subjects who qualify will go through clinical balance assessment and dynamic stability training. The older adults will be divided into any of the four groups -1) overground slip only training, 2) overground trip only training, 3) overground combined slip + trip training, or 4) control (single slip + single trip). For both overground slip/trip, all subjects' normal walking pattern and their recovery responses to slip/trip will be recorded with a motion tracking system (including videotaping) while they walk across an instrumented area along a straight path in the lab. A slip will be induced after a subject steps on a low-friction platform. A trip will be induced by introducing an obstacle device while the subject is walking, which consists of a hinged aluminum plate. At 12 months post-training session, the follow-up stability test will consist only of one slip and trip induced on the training side and contralateral side. Incidence of falls and physical activity will be monitored between training and re-test sessions through falls and activity monitoring-questionnaire to describe details of the falls.

ELIGIBILITY:
Inclusion Criteria:

* Community ambulators who use assistive device and are able to walk independently for 8m, healthy older adults between the age group of 60 to 90 years.
* Absence of any acute or chronic neurological, cardiopulmonary, musculoskeletal or systemic diagnosis.
* No recent major surgery (< 6 months) or hospitalization (< 3 months)
* Not on any sedative drugs.

Exclusion Criteria:

* Subjects will be excluded if they report presence of pain, osteoporosis or any medical conditions during telephone screening (see Telephone screening form). Also subjects will be excluded if they are on osteoporosis medication, and narcotics/opioids class of drugs under the sedative medications.
* Individuals classified as osteoporotic with heel bone density measurement with a T-score < -2 using an ultrasound device.
* Individuals with mild cognitive impairment (Mini-mental State Exam score < 25/30)
* Complain of shortness of breath or uncontrolled pain (> 3/10 on VAS) or pulse oxygen drops < 92% or are unable to achieve the age-specified minimal ambulation distance during 6 minute walk test.
* Subjects with body weight more than 250lbs.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in laboratory-induced falls | Baseline (1st novel slip, week 1), Immediate post-training (after repeated perturation training session, week 1 ) and at 12-month re-test (to determine long-term retention of training).
  Perturbation is induced successfully and safely to reproduce inadvertent falls in a protective laboratory environment. Falls will be measured by the amount of body weight supported by the full-body harness system and measured by a load cell attached to this system. Instability of the body's COM and poor limb support prior to touchdown of the recovery step account for 90~100% of subsequent falls (occurring ~500ms later) in both sit-to-stand-slip and in gait-slip, in the laboratory settings. Intervention consists of repeated perturbation training to induce a change in the laboratory induced falls immediately post-training and examine it's retention 12 months after the initial training session.
Real life falls | prospective post-training over next 12 months (total falls tracked and reported at 12 months post-training will be compared between groups)
  Real life falls are measured to determine if training effect can be translated into everyday real life setting.

SECONDARY OUTCOMES:
Stability gain (or loss) | Baseline (1st novel slip, week 1), Immediate post-training (after repeated perturation training session, week 1) and at 12-month re-test (to determine long-term retention of training).
  Stability is defined by both the position of a person's center-of-mass (COM) with respect to his or her base-of-support (BOS) and it's velocity.
Limb support gain (or loss) | Baseline (1st novel slip, week 1), Immediate post-training (after repeated perturation training session, week 1) and at 12-month re-test (to determine long-term retention of training).
  The inability to provide timely limb support due to insufficient amount of upward impulse generated from the ground reactive force can cause limb collapse, as characterized by the quotient of amount and rate of hip descent (Vhip/Zhip) measured from hip height and lead to an eventual fall.

CONTACTS AND LOCATIONS:
Overall Officials: Tanvi Bhatt, PhD PT, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhatt T, Wang Y, Wang S, Kannan L. Perturbation Training for Fall-Risk Reduction in Healthy Older Adults: Interference and Generalization to Opposing Novel Perturbations Post Intervention. Front Sports Act Living. 2021 Aug 16;3:697169. doi: 10.3389/fspor.2021.697169. eCollection 2021. PMID 34490424